CLINICAL TRIAL: NCT00022906
Title: Phase I, Dose-Escalation Study of Iodine-131 Anti-B1 Antibody For Patients With Previously Treated Non-Hodgkin's Lymphoma With More Than 25% Bone Marrow Involvement
Brief Title: Safety and Efficacy of Iodine-131 Anti-B1 Antibody for NHL Patients With Greater Than 25% Bone Marrow Involvement
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corixa Corporation (Industry)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-98-028
Record Dates: First submitted 2001-08-15; First posted 2001-08-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Radioimmunotherapy; Monoclonal Antibody; Corixa; Bexxar; Anti-B1 Antibody; Tositumomab; Iodine -131 Anti-B1 Antibody; Iodine I 131 Tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

INTERVENTIONS:
Drug: Iodine-131 Anti-B1 Antibody

SUMMARY:
The purpose of this study is to determine the proper dose, effectiveness, and safety of using Iodine-131 Anti-B1 Antibody for the treatment of patients with previously treated non-Hodgkin's lymphoma (NHL) who have greater than 25% bone marrow involvement with lymphoma.

DETAILED DESCRIPTION:
The primary endpoint is to determine the maximum tolerated dose of Iodine-131 Anti B-1 Antibody in patients with previously treated NHL having more than 25% bone marrow involvement with lymphoma. Secondary endpoints include assessment of response rate, duration of response, relapse-free survival, time to treatment failure, safety, and survival.

The dose escalation will be started at 45cGy and will be escalated in 10cGy increments until the maximum tolerated dose in reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed initial diagnosis of low-grade non-Hodgkin's B-cell lymphoma according to International Working Formulation (i.e., small lymphocytic [with or without plasmacytoid differentiation]; follicular small cleaved, or follicular, mixed small cleaved and large cell), or low-grade lymphoma that has transformed to a higher grade histology, or de novo follicular large cell lymphoma.
* Patients must have Ann Arbor Stage IV disease and greater than an average of 25% of the intratrabecular marrow space involved by NHL in bilateral bone marrow biopsy specimens as assessed microscopically at study entry. A unilateral bone marrow biopsy demonstrating greater than 50% involvement with NHL is also adequate for study entry.
* Patients must have been previously treated with chemotherapy and progressed on, failed to achieve an objective response on, or progressed after completion of their last chemotherapy.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen.
* Patients must have a performance status of at least 60% on the Karnofsky Performance Scale and an anticipated survival of at least 3 months.
* Patients must have an ANC greater than 1500 cells/mm3 and a platelet count greater than or equal to 150,000 cells/mm3 within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine less than 1.5 times the upper limit of normal) and hepatic function (defined as total bilirubin less than 1.5 times the upper limit of normal and AST less than 5 times the upper limit of normal) within 14 days of study entry.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be greater than or equal to 2 x 2 cm.

Exclusion Criteria:

* Patients with active obstructive hydronephrosis.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years. Patients who have been disease-free of another cancer for greater than 5 years must be carefully assessed at the time of study entry to rule out recurrent disease.
* Patients with known HIV infection.
* Patients who are HAMA positive.
* Patients with known brain or leptomeningeal metastases.
* Patients who have undergone therapy with either stem cell or bone marrow transplant.
* Patients who have received cytotoxic chemotherapy, immunosuppressants, or cytokine therapy within 4 weeks prior to study entry (6 weeks for nitrosourea compounds). The use of systemic steroids must be discontinued at least 1 week prior to study entry.
* Patients who are pregnant or breastfeeding. Patients of childbearing potential must undergo a serum pregnancy test within 7 days prior to study entry. Males and females must agree to use effective contraception for 6 months following the radioimmunotherapy dose.
* Patients with progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with more than 3500 cGy.
* Patients who are concurrently receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.
* Patients with active infection requiring IV anti-infectives at the time of study entry.
* Patients who have previously received radioimmunotherapy.
* Patients with de novo intermediate- or high-grade NHL, except for intermediate subtype of follicular large cell NHL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell Medical Center, New York, New York, United States